CLINICAL TRIAL: NCT01469195
Title: A Lead Rectangle to Lower the Radiation Exposure for Operators Who Uses Radial Approach in Coronary Procedures.
Brief Title: A Lead Rectangle to Lower the Operator's Radiation Exposure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: RAD410OSH
Record Dates: First submitted 2011-10-31; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Atherosclerosis; Coronary Occlusion; Coronary Artery Disease
Keywords: lead rectangle; radiation exposure; operators; radial approach; coronary procedures; percutaneous coronary intervention
MeSH Terms: conditions — Atherosclerosis; Coronary Occlusion; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A - No lead protection: Patients who are admitted for an elective percutaneous coronary intervention procedure ( or stable acute coronary syndrome patients) will be ask to participate in the study and sign an informed consent (see inclusions and exclusions).The Investigators will approach patients in whom a long procedure time and higher radiation exposure are anticipated (like patients with chronic total occlusion, heavily calcified or tortuous coronary arteries). In those, the fluoroscopy time on average, is longer than usual. In group A - no lead protection will be used.
- Group B plus lead protection: Patients who are admitted for an elective percutaneous coronary intervention procedure ( or stable acute coronary syndrome patients) will be ask to participate in the study and sign an informed consent (see inclusions and exclusions).The Investigators will approach patients in whom a long procedure time and higher radiation exposure are anticipated (like patients with chronic total occlusion, heavily calcified or tortuous coronary arteries). In those, the fluoroscopy time on average, is longer than usual. In group B - lead protection will be used from the umbilicus and down.

SUMMARY:
During fluoroscopic imaging, diagnostic information is carried in the primary beam. These high intensity X-rays are the chief hazard to the patient. Lower energy scattered radiation deviates in all directions from the patient. Despite typical precautions (i.e., hanging a lead shield between the patient and the operator), many operators will be exposed to high radiation dose (higher than the permitted 50 miliS per year), this long term radiation exposure may result in stochastic and deterministic effects. The purpose of this study was to test the hypothesis that a non disposable radiation protection drape (that will cover the lower part of the patient) could help minimize the radiation scattered from the patient to the operator. In a procedure done through the Radial approach, there is a large portion of the patients (from the umbilicus and down) that is a source of scatter radiation to the operator. This portion can be covered with a lead rectangle. A non disposable, lead drape of uniform thickness will be inserted into a sterile nylon bag and will be used during fluoroscopic and cineangiography coronary angioplasty procedures. The lead drapes will cover the femoral puncture site. The widths and length of the drape is 50-60cm and 100 cm respectively and was shown not to hinder the field of radiation needed for fluoroscopy and cineangiography. (The upper border of the lead is under the patient's umbilicus and was shown not to interfere with the radiation field needed for angiography or angioplasty).

The Investigators anticipate that the study will show a significant reduction in radiation exposure and hence reduce the radiation hazard to the operator.

DETAILED DESCRIPTION:
The Investigators tested the hypothesis on a Phantom that contain bones and tissue that simulate human tissue. The above phantom is used in the oncology department for testing radiation protocols delivered to patients. Those preliminary testing showed that a lead rectangle decreased significantly the radiation scattered towards the operators and personnel in the catheterization laboratory. In all chosen places whether 40 or 100 cm from the radiation beam - The Investigators detected a significant reduction in scattered radiation. The significant reduction in these experiments is attributed to the location the Investigators choose but also to the size of the lead drape 100 X60 cm which give a large area of protection. From simple geometric calculations it's understandable that the zone or volume of radiation protection become much larger further away from the lead rectangle.Patients who are admitted for an elective PCI procedure ( or stable ACS patients) will be ask to participate in the study and sign an informed consent. All the procedure will be as standard of care, after cleaning the right or left arm, and the groin a sterile towel will cover the groin, on top of the sterile towel the lead rectangle (that by itself will be inserted to a sterile nylon bag) will be put over to cover the area from the umbilicus and down.

(In case that the radial approach will fail and femoral approach will be needed, it is easy to remove the lead rectangle while keeping sterile field in the groin area). Few dosimeters will be used to assess radiation exposure, two underneath the lead apron, one on top, and two dosimeters for the operator (two detecting the radiation exposure in the neck area).

The Investigators will approach patients in whom a long procedure time and higher radiation exposure are anticipated (like patients with chronic total occlusion, heavily calcified or tortuous coronary arteries). In those, the fluoroscopy time on average, is longer than usual.

A total of 50 patients will be recruited (based on the Investigators preliminary radiation testing on the phantom and the results of Politi et al). In 25 patients a lead rectangle will be used on top of the regular protection (personal lead suit, leaded glass shield), in 25 patients only regular protection for the operators.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for an elective (non emergent) - radial access approach for coronary angioplasty.
* patients with angina pectoris or acute coronary syndrome, which are hemodynamically stable, will be included.
* Age 18-75.

Exclusion Criteria:

* Urgent/Emergent procedures (ST elevation myocardial infarction, suspected LM disease, low Ejection fraction <35%, patients in heart failure - NYHA class III, IV).
* Any situation that there is higher chance (over 10%) of switching to a femoral access approach (like weak radial pulse, low blood pressure <90 mmHg, failed radial access in the past) .
* Significant valve disease like; severe aortic stenosis, severe mitral regurgitation.
* Pregnancy or women in child bearing age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective or acute coronary syndrome patients who go through percutaneous coronary intervention at one tertiary centre
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
scattered radiation reduction with lead rectangle protection Vs. no protection at distance of 40-100 cm from the radiation beam | Outcome measure is assessed same day immediately after the procedure (recording the dose of radiation detected by the dosimeters) participants will be followed for the duration of hospital stay, an expected average of 2-4 days.
  The Investigators will use "Inlight" (Landauer) dosimeters that are sensitive and can be read over and over to give the differences in scattered radiation, (with or without the lead rectangle). these dosimeters will be read Immediately at the end of the procedure. The investigators will look for the difference in the readings between patients that had the lead rectangle on to patients without the lead rectangle.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Strauss, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre, Schulich Heart program Devision of Cardiology Toronto Ontario, Canada
Locations (1):
- Sunnybrook health sciences centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Politi L, Biondi-Zoccai G, Nocetti L, Costi T, Monopoli D, Rossi R, Sgura F, Modena MG, Sangiorgi GM. Reduction of scatter radiation during transradial percutaneous coronary angiography: a randomized trial using a lead-free radiation shield. Catheter Cardiovasc Interv. 2012 Jan 1;79(1):97-102. doi: 10.1002/ccd.22947. Epub 2011 Apr 25. PMID 21520391